CLINICAL TRIAL: NCT04451837
Title: Semaglutide and Dapagliflozin in Diabetic Patients With Different Pathophysiology
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIAB1
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — semaglutide; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- semaglutide (Active Comparator): Patients randomized to add semaglutide (Ozempic) will receive injection training at the study site and inject 0.25 mg subcutaneously once weekly during the first four weeks, followed by 0.5 mg weekly for the subsequent four weeks and finally 1.0 mg weekly throughout the study.
  Interventions: Drug: Semaglutide
- dapagliflozin (Active Comparator): Those randomized to dapagliflozin will receive 10 mg orally once daily in addition to metformin.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Semaglutide — Ozempic s.c. once weekly for 6 months
  Other Names: Ozempic
  Arms: semaglutide
Drug: Dapagliflozin — Forxiga 10 mg p.o. once daily for 6 months
  Other Names: Forxiga
  Arms: dapagliflozin

SUMMARY:
Current anti-diabetic treatment fails to stop the progressive course of the disease. Recent studies have revealed a surprisingly high variability in the diabetic phenotype. The investigators propose that anti-diabetic treatment should ideally target the underlying pathophysiology of each individual patient. The investigators will therefore test whether the effect of two approved anti-diabetic drugs differs between individuals at different ends of the pathophysiological spectrum: 1) patients with poor insulin secretion, here termed SIDD and 2) patients with high insulin resistance, here termed SIRD. The study may open up a new avenue for more precise treatment of diabetic patients that would be of immediate clinical relevance.

DETAILED DESCRIPTION:
The trial is a clinical phase II study that will be randomized and open-label with fixed stratification variables (SIDD and SIRD) to analyze if the response to anti-diabetic drugs differs between patients with distinct pathophysiology, as captured by SIDD and SIRD. The compounds used are semaglutide and dapagliflozin, which will be randomized to patients of each subgroup using a parallel group design.

The clusters (SIDD and SIRD) will be used as a practical tool to distinguish individuals who are at different ends of the pathophysiological spectrum.

The investigators will recruit 200 patients from the ANDIS registry with HbA1c ≥42 mmol/mol on metformin monotherapy. Half of them will have SIDD and half will have SIRD characteristics. The patients will be randomized (open-label) to receive semaglutide or dapagliflozin for six months in addition to metformin.

The investigators will recruit participants on metformin monotherapy with stable dose for the last three months. Metformin dose at inclusion (as prescribed by their regular physician) is maintained throughout the study; the investigatorswill correct for metformin dose in the analyses. Patients randomized to add semaglutide will receive injection training at the study site and inject 0.25 mg subcutaneously once weekly during the first four weeks, followed by 0.5 mg weekly for the subsequent four weeks and finally 1.0 mg weekly throughout the study. Those randomized to dapagliflozin will receive 10 mg orally once daily in addition to metformin. The participants will attend a screening visit followed by three study visits at 0, 3, 6 months. At the first and last study visit they will undergo an OGTT. HbA1c will be measured at all study visits.

ELIGIBILITY:
Inclusion Criteria:

* • Diabetes mellitus based on prior documentation or treatment with anti-hyperglycemic medication or diagnosed according to the WHO criteria (random plasma glucose >11.1 mmol/L or fasting glucose >7.0 mmol/L or HbA1C ≥6.5%) and disease characteristics typical for SIDD or SIRD according to the ANDIS clustering

  * Ongoing metformin therapy with constant dose the last three months
  * Age 18 years or above
  * HbA1c ≥42 and <91 mmol/mol
  * Women who are not postmenopausal and who have not undergone surgical sterilization must have no current pregnancy, which will be assessed by pregnancy test, must take precautions to avoid pregnancy throughout the study and for 4 weeks after intake of the last dose and must be willing to use highly effective birth control methods. Methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods.
  * Willingness to take injectable and oral medication
  * Written informed consent

Exclusion Criteria:

* • Type 1 diabetes, LADA, MODY, secondary diabetes or history of diabetic ketoacidosis

  * Anti-diabetic treatment other than metformin within 90 days prior to randomization or changed metformin dose within 90 days prior to randomization
  * Known acute cardiovascular event, e.g. transient ischemic attack, stroke, acute coronary syndrome, decompensated heart failure, coronary by-pass surgery or other coronary vessel intervention within 90 days prior to screening.
  * Heart failure NYHA class IV
  * History of acute or chronic pancreatitis
  * Known liver cirrhosis
  * Blood pressure above 170/110 mm Hg
  * A level of aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT), ALP or bilirubin of more than three times the upper limit of the normal range
  * Current chronic daily treatment with an oral steroid at a dose equivalent to oral prednisolone ≥10 mg (e.g., betamethasone ≥1.2 mg, dexamethasone ≥1.5 mg, hydrocortisone ≥40 mg)
  * Pregnancy or breast-feeding
  * Known galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.
  * Estimated glomerular filtration rate <45 ml/min/1,73 m2 or unstable or rapidly progressing renal disease
  * Participant unable to understand the study information herself or himself
  * Involvement in the planning and/or conduct of the study
  * Participation in other clinical trial which may affect the outcome of the present study
  * Any condition or treatment that in the judgment of the investigator makes it difficult or unsafe to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hba1c | 6 months
  The primary endpoint will be the intraindividual change of HbA1c in response to semaglutide or dapagliflozin relative to baseline in the two patient groups.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Rosengren, Principal Investigator — Region Skåne
Locations (1):
- Anders Rosengrentest, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dwibedi C, Ekstrom O, Brandt J, Adiels M, Franzen S, Abrahamsson B, Rosengren AH. Randomized open-label trial of semaglutide and dapagliflozin in patients with type 2 diabetes of different pathophysiology. Nat Metab. 2024 Jan;6(1):50-60. doi: 10.1038/s42255-023-00943-3. Epub 2024 Jan 4. PMID 38177805